CLINICAL TRIAL: NCT03229863
Title: The Infant MiND Study: An Examination of Infants' Microbiome, Nutrition, and Development Study.
Brief Title: An Examination of Infants' Microbiome, Nutrition, and Development Study.
Acronym: IMiND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: UC Davis Foods for Health Institute (Unknown); Mengniu Dairy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 919505
Record Dates: First submitted 2017-07-07; First posted 2017-07-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Microbial Colonization; Infant Development
Keywords: Breastfeeding; First foods
MeSH Terms: conditions — Communicable Diseases; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This study is designed as a combined randomized, crossover interventional and observational trial. At the start of the study, infants will enter a 7-day lead-in period to establish gut microbiome and GI tolerability baselines. After the 7-day lead-in period, infants will be randomized into one of two feeding arms comprised of two commercially available baby foods: sweet potato (SP) (Plum Organics, Just Sweet Potato) and pears (P) (Earth's Best, First Pears). The first food, either sweet potato or pears, will be consumed for 7 days followed by a 4-day washout period of exclusive breast milk before initiating the alternate 7-day feeding arm of pears or sweet potato, respectively. The second feeding arm will be followed by an additional 4-day washout period of exclusive breast milk before the introduction of any other solid foods. Once the first month of the study is complete, infants will enter an observational phase for the remainder of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweet Potatos (Experimental): Infants will consume commercially available baby food sweet potato (SP) (Plum Organics, Just Sweet Potato) for 7 days followed by a 4 day washout period of exclusive breast milk. Participants will be instructed to offer 1-2 tablespoons of sweet potato to their infant at least three times per day for seven days in a row.
  Interventions: Other: Sweet Potatos
- Pears (Experimental): Infants will consume commercially available baby food pear (P) (Earth's Best, First Pears) for 7 days followed by a 4 day washout period of exclusive breast milk. Participants will be instructed to offer 1-2 tablespoons of pears to their infant at least three times per day for seven days in a row.
  Interventions: Other: Pears

INTERVENTIONS:
Other: Sweet Potatos — Plum Organics, Just Sweet Potato
  Arms: Sweet Potatos
Other: Pears — Earth's Best, First Pears
  Arms: Pears

SUMMARY:
This study is examining the relationship between infant nutrition, gut health, and development. The fecal microbiota changes and develops, in large part due to the food that infants eat. These changes are important for many aspects of development. This study is designed to examine how the fecal microbiota changes when exclusively breastfed infants are first introduced to solid food, and how changes of the fecal microbiota are related to other aspects of development.

DETAILED DESCRIPTION:
The purpose of this study is to determine: 1) how the gut bacteria of exclusively breastfed infants changes in response to ingesting solid foods; 2) how infant cognition develops in response to ingesting solid foods; and 3) the relationship between infant gut bacteria and infant cognition during the first year of life.

This study is designed to determine how specific complex carbohydrates in commonly used first foods encourage the growth of different bacteria in the infant gut. The two foods used in this study are commercially-available sweet potato (Plum Organics) and pear (Earth's Best). These two foods have been chosen because they differ substantially from each other in their carbohydrate composition. For example, sweet potato is mostly made up of starch which is digestible and pear is made up of other types of sugars found in fruits and vegetables that are not digestible and may have "prebiotic" effects (food for good bacteria in the gut). Thus, the use of these two foods could provide a good contrast for comparing how gut bacteria respond to different carbohydrate compositions during complementary feeding.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 21 to 45 years who have delivered a healthy single infant by vaginal delivery and their infants, age 4 to 7.5 months;
* Infants who are developmentally ready for solids;
* Generally healthy women and infants;
* Mothers who plan to exclusively (without solids or infant formula) breastfeed (at the breast or feed breast milk by bottle) their infants for at least 5 months of age and plan to continue to breastfeed with solids and/or infant formula until 12 months of age;
* Mothers who are willing to either use their own breast pump, or hand-express, or use a manual pump provided by the study to collect milk samples;
* Mothers who are willing to refrain from feeding their infants infant formula, non-study solid foods; probiotic or iron supplements (confounding variables of the intestinal microbiome) before the end of the feeding intervention period;
* Term infants born >37 weeks gestation;
* Mother-infant pairs who live within a 20-mile radius from University of California, Davis campus in Davis, California (includes Woodland, Vacaville, Dixon and surrounding areas) or within a 20-mile radius of the University of California, Davis Medical Center (UCDMC) (2221 Stockton Blvd, Sacramento, CA 95817).

Exclusion Criteria:

* Infants with any GI tract abnormalities;
* Infants born by cesarean section;
* Family history of immunodeficiency syndrome(s);
* Multiple infants born to one mother at the same time (no twins, triplets, etc.);
* Infants born with medical complications such as: respiratory distress syndrome, birth defects, and infection;
* Mothers diagnosed with any metabolic or endocrine, liver, kidney disease, any autoimmune disease, cirrhosis, hepatitis C, HIV, AIDS, cancer, obesity (pre-pregnancy BMI >34.9), polycystic ovary syndrome (PCOS), celiac disease, Crohn's disease, heart disease, hyper- or hypothyroidism, hyper- or hypotension (including pre-eclampsia), type 1 or type 2 diabetes.
* Mothers who smoked cigarettes less than one month before becoming pregnant, during pregnancy, and currently or mothers who plan to initiate smoking during the study duration;
* Infants who have taken antibiotics within the past 4 weeks;
* Infants who have taken iron supplements within the past 4 weeks;
* Infants who have consumed infant formula in the past 4 weeks;
* Infants who have consumed infant formula more than 10 days between birth and 4 weeks prior to screening;
* Infants who have consumed any solids;
* Mothers who plan to feed infants solids before 5 months of age;
* Mothers who plan to administer any probiotics to infants throughout the feeding intervention period (first 18 days of the study);
* Infants who have consumed probiotics containing Bifidobacterium within the past 4 weeks or other probiotics within the past 7 days;
* Mothers who live in more than one location (should only live in one house to ensure samples are correctly collected and stored);
* Infants who have hypotonia,
* Infants who have been diagnosed with any medical or nutritional condition that would require iron supplementation.
* Infants who on average pass less than one stool per week.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Infant fecal microbiota composition | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The difference in the relative abundance of the infant fecal microbiome at the order level (top 22 taxonomic orders with abundance expressed as both on log10 scale and a percent of total bacteria) between baseline and post-complementary food intake for each intervention arm (sweet potato vs. pear).
Infant fecal microbial diversity | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The difference in the infant fecal microbial diversity and microbial function between baseline and post-complementary food intake for each arm (sweet potato vs. pear)
Incidence of Adverse Events and Treatments | Baseline-days 180
  Incidence of gastrointestinal symptoms (discomfort passing bowel movements, vomiting, constipation, colic or irritability), illnesses, health care visits for sickness, high fevers, antibiotic and medication use.

SECONDARY OUTCOMES:
Dietary composition | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between the relative abundance of the infant fecal microbiome and function, and food glycan composition.
Infant cognition | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between the relative abundance of the infant fecal microbiome, microbial diversity and function, and infant cognition measured at 6, 8 and 12 months of age
Infant sleep | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between the relative abundance of the infant fecal microbiome, microbial diversity and function, and infant sleep, activity and vocalizations measured throughout the study period.
Maternal secretor status and infant fecal microbiota | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between maternal secretor status (via measurement of human milk oligosaccharides in breast milk) and the relative abundance of the infant fecal microbiome, microbial diversity and function before, during and after introduction of complementary foods.
Infant secretor status and fecal microbiota | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between infant secretor status (via measurement of oligosaccharides in saliva) the relative abundance of the infant fecal microbiome, microbial diversity and function before, during and after introduction of complementary foods.
Maternal and infant fecal microbiota | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The relationship between maternal and infant fecal microbiome.
Infant fecal human milk oligosaccharide concentrations | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  The change in infant fecal human milk oligosaccharide concentrations before, during and after introduction of complementary foods.
Infant weight | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  Determine the relationship between infant weight and the relative abundance of the infant fecal microbiome, microbial diversity and function before, during and after introduction of complementary foods
Human milk metabolomics | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  Determine the relationship between human milk metabolomics (metabolites, fatty acids, proteins) and the infant fecal microbiome.
Fecal metabolomics | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  Determine the relationship between fecal metabolites (metabolites, fatty acids, proteins) and fecal microbiome.
Infant gastrointestinal function | Change from baseline, days 14, 19, 25, 29, 60, 90, 120, 150, 180
  Change in GI function as a means to monitor tolerability before, during and after introduction of complementary foods (through the measurement of fecal inflammatory mediators, GI barrier function markers and fecal LPS).
Glycosidic linkages | Change from baseline to day 29
  Evaluate the glycosidic linkages in interventional foods and the infant fecal microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smilowitz, PhD, Principal Investigator — University of California, Davis; Lisa Oakes, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

REFERENCES:
- [Background] Hoskin-Parr L, Teyhan A, Blocker A, Henderson AJ. Antibiotic exposure in the first two years of life and development of asthma and other allergic diseases by 7.5 yr: a dose-dependent relationship. Pediatr Allergy Immunol. 2013 Dec;24(8):762-71. doi: 10.1111/pai.12153. Epub 2013 Dec 2. PMID 24299467
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Makino H, Kushiro A, Ishikawa E, Muylaert D, Kubota H, Sakai T, Oishi K, Martin R, Ben Amor K, Oozeer R, Knol J, Tanaka R. Transmission of intestinal Bifidobacterium longum subsp. longum strains from mother to infant, determined by multilocus sequencing typing and amplified fragment length polymorphism. Appl Environ Microbiol. 2011 Oct;77(19):6788-93. doi: 10.1128/AEM.05346-11. Epub 2011 Aug 5. PMID 21821739
- [Background] Backhed F, Roswall J, Peng Y, Feng Q, Jia H, Kovatcheva-Datchary P, Li Y, Xia Y, Xie H, Zhong H, Khan MT, Zhang J, Li J, Xiao L, Al-Aama J, Zhang D, Lee YS, Kotowska D, Colding C, Tremaroli V, Yin Y, Bergman S, Xu X, Madsen L, Kristiansen K, Dahlgren J, Wang J. Dynamics and Stabilization of the Human Gut Microbiome during the First Year of Life. Cell Host Microbe. 2015 May 13;17(5):690-703. doi: 10.1016/j.chom.2015.04.004. PMID 25974306
- [Background] Penders J, Thijs C, Vink C, Stelma FF, Snijders B, Kummeling I, van den Brandt PA, Stobberingh EE. Factors influencing the composition of the intestinal microbiota in early infancy. Pediatrics. 2006 Aug;118(2):511-21. doi: 10.1542/peds.2005-2824. PMID 16882802
- [Background] Bezirtzoglou E, Tsiotsias A, Welling GW. Microbiota profile in feces of breast- and formula-fed newborns by using fluorescence in situ hybridization (FISH). Anaerobe. 2011 Dec;17(6):478-82. doi: 10.1016/j.anaerobe.2011.03.009. Epub 2011 Apr 8. PMID 21497661
- [Background] Mitsuoka T, Kaneuchi C. Ecology of the bifidobacteria. Am J Clin Nutr. 1977 Nov;30(11):1799-810. doi: 10.1093/ajcn/30.11.1799. No abstract available. PMID 920640
- [Background] Sela DA, Chapman J, Adeuya A, Kim JH, Chen F, Whitehead TR, Lapidus A, Rokhsar DS, Lebrilla CB, German JB, Price NP, Richardson PM, Mills DA. The genome sequence of Bifidobacterium longum subsp. infantis reveals adaptations for milk utilization within the infant microbiome. Proc Natl Acad Sci U S A. 2008 Dec 2;105(48):18964-9. doi: 10.1073/pnas.0809584105. Epub 2008 Nov 24. PMID 19033196
- [Background] Sela DA, Garrido D, Lerno L, Wu S, Tan K, Eom HJ, Joachimiak A, Lebrilla CB, Mills DA. Bifidobacterium longum subsp. infantis ATCC 15697 alpha-fucosidases are active on fucosylated human milk oligosaccharides. Appl Environ Microbiol. 2012 Feb;78(3):795-803. doi: 10.1128/AEM.06762-11. Epub 2011 Dec 2. PMID 22138995
- [Background] Sela DA, Li Y, Lerno L, Wu S, Marcobal AM, German JB, Chen X, Lebrilla CB, Mills DA. An infant-associated bacterial commensal utilizes breast milk sialyloligosaccharides. J Biol Chem. 2011 Apr 8;286(14):11909-18. doi: 10.1074/jbc.M110.193359. Epub 2011 Feb 2. PMID 21288901
- [Background] Garrido D, Kim JH, German JB, Raybould HE, Mills DA. Oligosaccharide binding proteins from Bifidobacterium longum subsp. infantis reveal a preference for host glycans. PLoS One. 2011 Mar 15;6(3):e17315. doi: 10.1371/journal.pone.0017315. PMID 21423604
- [Background] LoCascio RG, Ninonuevo MR, Freeman SL, Sela DA, Grimm R, Lebrilla CB, Mills DA, German JB. Glycoprofiling of bifidobacterial consumption of human milk oligosaccharides demonstrates strain specific, preferential consumption of small chain glycans secreted in early human lactation. J Agric Food Chem. 2007 Oct 31;55(22):8914-9. doi: 10.1021/jf0710480. Epub 2007 Oct 5. PMID 17915960
- [Background] Krebs NF, Sherlock LG, Westcott J, Culbertson D, Hambidge KM, Feazel LM, Robertson CE, Frank DN. Effects of different complementary feeding regimens on iron status and enteric microbiota in breastfed infants. J Pediatr. 2013 Aug;163(2):416-23. doi: 10.1016/j.jpeds.2013.01.024. Epub 2013 Feb 26. PMID 23452586
- [Background] Arumugam M, Raes J, Pelletier E, Le Paslier D, Yamada T, Mende DR, Fernandes GR, Tap J, Bruls T, Batto JM, Bertalan M, Borruel N, Casellas F, Fernandez L, Gautier L, Hansen T, Hattori M, Hayashi T, Kleerebezem M, Kurokawa K, Leclerc M, Levenez F, Manichanh C, Nielsen HB, Nielsen T, Pons N, Poulain J, Qin J, Sicheritz-Ponten T, Tims S, Torrents D, Ugarte E, Zoetendal EG, Wang J, Guarner F, Pedersen O, de Vos WM, Brunak S, Dore J; MetaHIT Consortium; Antolin M, Artiguenave F, Blottiere HM, Almeida M, Brechot C, Cara C, Chervaux C, Cultrone A, Delorme C, Denariaz G, Dervyn R, Foerstner KU, Friss C, van de Guchte M, Guedon E, Haimet F, Huber W, van Hylckama-Vlieg J, Jamet A, Juste C, Kaci G, Knol J, Lakhdari O, Layec S, Le Roux K, Maguin E, Merieux A, Melo Minardi R, M'rini C, Muller J, Oozeer R, Parkhill J, Renault P, Rescigno M, Sanchez N, Sunagawa S, Torrejon A, Turner K, Vandemeulebrouck G, Varela E, Winogradsky Y, Zeller G, Weissenbach J, Ehrlich SD, Bork P. Enterotypes of the human gut microbiome. Nature. 2011 May 12;473(7346):174-80. doi: 10.1038/nature09944. Epub 2011 Apr 20. PMID 21508958
- [Background] Davis LM, Martinez I, Walter J, Hutkins R. A dose dependent impact of prebiotic galactooligosaccharides on the intestinal microbiota of healthy adults. Int J Food Microbiol. 2010 Dec 15;144(2):285-92. doi: 10.1016/j.ijfoodmicro.2010.10.007. Epub 2010 Oct 14. PMID 21059476
- [Background] Faith JJ, Guruge JL, Charbonneau M, Subramanian S, Seedorf H, Goodman AL, Clemente JC, Knight R, Heath AC, Leibel RL, Rosenbaum M, Gordon JI. The long-term stability of the human gut microbiota. Science. 2013 Jul 5;341(6141):1237439. doi: 10.1126/science.1237439. PMID 23828941
- [Background] Martinez I, Muller CE, Walter J. Long-term temporal analysis of the human fecal microbiota revealed a stable core of dominant bacterial species. PLoS One. 2013 Jul 16;8(7):e69621. doi: 10.1371/journal.pone.0069621. Print 2013. PMID 23874976
- [Background] de Theije CG, Wopereis H, Ramadan M, van Eijndthoven T, Lambert J, Knol J, Garssen J, Kraneveld AD, Oozeer R. Altered gut microbiota and activity in a murine model of autism spectrum disorders. Brain Behav Immun. 2014 Mar;37:197-206. doi: 10.1016/j.bbi.2013.12.005. Epub 2013 Dec 11. PMID 24333160
- [Background] Foster JA, McVey Neufeld KA. Gut-brain axis: how the microbiome influences anxiety and depression. Trends Neurosci. 2013 May;36(5):305-12. doi: 10.1016/j.tins.2013.01.005. Epub 2013 Feb 4. PMID 23384445
- [Background] Song Y, Liu C, Finegold SM. Real-time PCR quantitation of clostridia in feces of autistic children. Appl Environ Microbiol. 2004 Nov;70(11):6459-65. doi: 10.1128/AEM.70.11.6459-6465.2004. PMID 15528506
- [Background] Wang L, Christophersen CT, Sorich MJ, Gerber JP, Angley MT, Conlon MA. Low relative abundances of the mucolytic bacterium Akkermansia muciniphila and Bifidobacterium spp. in feces of children with autism. Appl Environ Microbiol. 2011 Sep;77(18):6718-21. doi: 10.1128/AEM.05212-11. Epub 2011 Jul 22. PMID 21784919
- [Background] Diaz Heijtz R, Wang S, Anuar F, Qian Y, Bjorkholm B, Samuelsson A, Hibberd ML, Forssberg H, Pettersson S. Normal gut microbiota modulates brain development and behavior. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3047-52. doi: 10.1073/pnas.1010529108. Epub 2011 Jan 31. PMID 21282636
- [Background] Collins SM, Surette M, Bercik P. The interplay between the intestinal microbiota and the brain. Nat Rev Microbiol. 2012 Nov;10(11):735-42. doi: 10.1038/nrmicro2876. Epub 2012 Sep 24. PMID 23000955
- [Background] Borre YE, O'Keeffe GW, Clarke G, Stanton C, Dinan TG, Cryan JF. Microbiota and neurodevelopmental windows: implications for brain disorders. Trends Mol Med. 2014 Sep;20(9):509-18. doi: 10.1016/j.molmed.2014.05.002. Epub 2014 Jun 20. PMID 24956966
- [Background] Totten SM, Zivkovic AM, Wu S, Ngyuen U, Freeman SL, Ruhaak LR, Darboe MK, German JB, Prentice AM, Lebrilla CB. Comprehensive profiles of human milk oligosaccharides yield highly sensitive and specific markers for determining secretor status in lactating mothers. J Proteome Res. 2012 Dec 7;11(12):6124-33. doi: 10.1021/pr300769g. Epub 2012 Nov 19. PMID 23140396
- [Background] Tao N, DePeters EJ, Freeman S, German JB, Grimm R, Lebrilla CB. Bovine milk glycome. J Dairy Sci. 2008 Oct;91(10):3768-78. doi: 10.3168/jds.2008-1305. PMID 18832198
- [Background] Tao N, DePeters EJ, German JB, Grimm R, Lebrilla CB. Variations in bovine milk oligosaccharides during early and middle lactation stages analyzed by high-performance liquid chromatography-chip/mass spectrometry. J Dairy Sci. 2009 Jul;92(7):2991-3001. doi: 10.3168/jds.2008-1642. PMID 19528576
- [Background] Vatanen T, Kostic AD, d'Hennezel E, Siljander H, Franzosa EA, Yassour M, Kolde R, Vlamakis H, Arthur TD, Hamalainen AM, Peet A, Tillmann V, Uibo R, Mokurov S, Dorshakova N, Ilonen J, Virtanen SM, Szabo SJ, Porter JA, Lahdesmaki H, Huttenhower C, Gevers D, Cullen TW, Knip M; DIABIMMUNE Study Group; Xavier RJ. Variation in Microbiome LPS Immunogenicity Contributes to Autoimmunity in Humans. Cell. 2016 May 5;165(4):842-53. doi: 10.1016/j.cell.2016.04.007. Epub 2016 Apr 28. PMID 27133167
- [Background] Rotmistrovsky, K. and R. Agarwala, BMTagger: Best Match Tagger for removing human reads from metagenomics datasets. 2011.
- [Background] Schmieder R, Edwards R. Fast identification and removal of sequence contamination from genomic and metagenomic datasets. PLoS One. 2011 Mar 9;6(3):e17288. doi: 10.1371/journal.pone.0017288. PMID 21408061
- [Background] Ames SK, Gardner SN, Marti JM, Slezak TR, Gokhale MB, Allen JE. Using populations of human and microbial genomes for organism detection in metagenomes. Genome Res. 2015 Jul;25(7):1056-67. doi: 10.1101/gr.184879.114. Epub 2015 Apr 29. PMID 25926546
- [Background] Kleinman RE. American Academy of Pediatrics recommendations for complementary feeding. Pediatrics. 2000 Nov;106(5):1274. No abstract available. PMID 11061819
- See also: Learn more or sign up for the study here! — https://studypages.com/s/an-examination-of-infants-microbiome-nutrition-and-development-study-123299/